CLINICAL TRIAL: NCT05042947
Title: Feasibility of a New Ligation Using the Double-loop Clips Technique Versus Traditional Techniques in the Treatment of Large Wounds After Endoscopic Resection: a Prospective Randomized Controlled Study
Brief Title: A New Ligation Using the Double-loop Clips Technique Versus Traditional Techniques in the Treatment of Large Wounds After Endoscopic Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLCT-1.0
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Polyps; Closure; Delay
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DLCT (Experimental): After finding polyps that meet the inclusion criteria, the surgical method for resection was selected according to the operator's preferences, and the experimental group used double-loop coil clamp technology to treat the wound.
  Interventions: Device: double-loop clips
- Traditional technology (Active Comparator): After finding polyps that meet the inclusion criteria, the surgical method for resection was selected according to the operator's preferences.The control group used the traditional hemostatic clip technique to treat the wound
  Interventions: Device: Titanium Clip

INTERVENTIONS:
Device: double-loop clips — a new ligation method using the double-loop clips (D-L clips) technique
  Arms: DLCT
Device: Titanium Clip — the Titanium Clip
  Other Names: Traditional technology
  Arms: Traditional technology

SUMMARY:
Studies have shown that postoperative inflammation can be relieved by clipping the wound, and can reduce the bleeding rate and perforation rate.Scholars at home and abroad have proposed the use of adhesives and circular surgical lines to clamp the wound.In 2019, Satoshi Abiko and others proposed the use of double-loop clips technology to clamp the wound, and make double-loop clips of appropriate length outside the body.Therefore, our study is a prospective randomized controlled study to explore whether the double-loop clips technique is safe and effective for larger wounds in daily clinical work.

ELIGIBILITY:
Inclusion Criteria:

* Patients with wounds larger than 20mm
* Patients aged 18 to 75 years old

Exclusion Criteria:

* Have a serious medical condition, such as heart failure, acute liver failure, severe kidney disease (dialysis or predialysis patients) or New York heart association class iii-iv.
* Pregnant or breastfeeding.
* Allergy or intolerance to any study drug.
* Patients who have taken anticoagulant drugs (aspirin, clopidogrel, etc.) in the past week but are contraindicated for endoscopic polyp treatment.
* Other imaging findings suggest patients with advanced cancer.
* Patients with severe gastrointestinal diseases, such as intestinal obstruction or perforation, active ulcerative colitis, toxic colitis, and toxic megacolon

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
complete closure rate | 1 hour
  Main outcome was complete clip closure of the mucosal resection defect. The defect was considered completely closed when there was no remaining visible mucosal defect and clips were <1cm apart.

SECONDARY OUTCOMES:
Operating time | 1 hour
  The time from when the first clip is hit until it is completely closed
Closing speed | 1 hour
  Resection area divided by clamping time

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China